CLINICAL TRIAL: NCT05343195
Title: Effect of Task-Specific Exercise on Balance and Leg Function in Patients After Total Hip Replacement
Brief Title: Balance and Leg Function After Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LithuanianSportsU-9
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Hip Injuries; Coxarthrosis; Hip Replacement
Keywords: balance; hip function; hip replacement; elderly; physical functioning
MeSH Terms: conditions — Hip Injuries; Osteoarthritis, Hip

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Conventional physiotherapy was applied 5 days/ week, 30 min session, in total 18 days.
  Exercise program:
  * 1-2 week: 20 min. of active exercise in lying position (e.g.: hip flexion, extension, abduction) with the goal to improve hip range of motions, strengthen muscles. Various equipment was used (slippery base, elastic bands, foam roller, gymnastic ball etc.). + gait training exercise within the bars (10 min);
  * 3 week: 20 min. of active exercise in lying position + stationary bicycle / treadmill (10 min).
  Interventions: Other: Control
- Task oriented exercise group (Experimental): Task oriented exercise program was applied 5 days/ week, 30 min session, in total 18 days.
  Exercise program included:
  * 1 week: active exercise in lying position (15 min) + task-oriented exercise (15 min);
  * 2 week: active exercise in lying position (10 min) + task-oriented exercise (20 min);
  * 3 week: stationary bicycle / treadmill (10 min) + task-oriented exercise (20 min).
  Task oriented exercise included:
  * walking backwards, sideways, high kneels (on the instable bases);
  * walking with alternate speed (physiotherapist give the instruction when to walk faster / slower);
  * Sit and stand from the chair (standing up to reach for the ball held by the physiotherapist);
  * step onto the step (after stepping to reach the ball held by the physiotherapist);
  * walk with the obstacles (obstacle course);
  * Catch and throw the ball while standing on an unstable base.
  Interventions: Other: Task-oriented exercise

INTERVENTIONS:
Other: Task-oriented exercise — Task-oriented exercise program for patients after total hip replacement.
  Arms: Task oriented exercise group
Other: Control — Control intervention: conventional physiotherapy after hip replacement
  Arms: Control group

SUMMARY:
Task-oriented leg exercise are commonly used after joint surgeries in various hip pathologies. Based on this theory, it was hypothesized that task-oriented exercise without conventional physiotherapy can have better result in recovery of balance and leg function than with a conventional post-hip physiotherapy program after hip replacement surgery. The aim of the study was to determine the effect of task-oriented exercise on balance and leg function after total hip replacement.

DETAILED DESCRIPTION:
Study included 40 subjects. All subjects were randomly divided into control and intervention groups. VAS scale was used to assess the pain, hip range of motion were measured using a goniometer, strength of the muscles was assessed on the Oxford 5 point scale, leg function was evaluated with modified Harris hip scale, Abili balance analyzer was used to assess static balance and Berg balance scale was used to measure dynamic balance. Intervention duration was 18 days.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 40;
* Hip coxarthrosis;
* Hip total replacement;
* Posterior incision;
* Surgery performed no more than 1 week ago;
* Ability to comprehend and execute the tasks.

Exclusion Criteria:

* Revision surgery;
* Surgery intervention for other reasons (fracture, arthritis);
* Severe cardiovascular disease;
* Vestibular disorders;
* Vision disorders;
* Proprioception disorders;
* Neurological disorders.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline Pain at 18 days | Baseline and after 18 days
  was evaluated using the Visual Analogue Pain Scale (VAS). Participants were asked to report "current" pain intensity. A higher score indicates greater pain intensity: no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), and severe pain (75- 100 mm).
Change from baseline Hip range of motions at 18 days | Baseline and after 18 days
  Using goniometer the range of hip motions were evaluated: flexion, extension, abduction. Each motion was measured three times and averaged value was used.
Change from baseline Hip Muscle Strength at 18 days | Baseline and after 18 days
  The muscle strength of hip flexion, extension, and abduction was evaluated using manual muscle testing technique (Oxford 5 point scale).
Change from baseline Leg Function at 18 days | Baseline and after 18 days
  To evaluate the function of leg after hip replacement surgery the modified Harris Hip Score (mHHS) was used. MHHS is reliable and valid tool to evaluate leg function after hip replacement and to monitor the leg function during recovery. The questionnaire was completed by a physiotherapist together with the patient. This questionnaire consists of 8 questions / topics, where each answer has a score:
  * Pain description (maximum 44 points);
  * Limping (max 11 points);
  * Assistive devices (max 11 points);
  * Walking distance (max 11 points);
  * Stair climbing (max 4 points);
  * Putting on shoes/socks (max 4 points);
  * Sitting (max 5 points);
  * Using public transport (1 point). The higher the score, the better the leg function. The maximum number of points is 91.
Change from baseline Dynamic Balance at 18 days | Baseline and after 18 days
  Dynamic Balance was assessed using the Berg Balance Scale (BBS). This scale is used to assess the subjects' imbalance in 14 different tasks, where each task is scored on a scale from 0 (does not perform at all) to 4 (performs excellent). The higher the score, the better the balance, with a maximum score of 56.
Change from baseline Static Balance at 18 days | Baseline and after 18 days
  Static Balance was assessed using the "Abili balance analyzer system". Abili balance analyzer is a platform that can be adapted for both patient testing and training. The Abili analyzer system consists of two parts: the Abili analyzer platform and the Balance trainer app. The Abili analyzer platform plate moves in a horizontal plane, making it safe to use for patients of all capacities. Thus, using this balance platform, three levels of difficulty can be selected: light, medium and advanced, as well as the handles are adjustable according to the patient's height. After three tests, the gadget calculates a total stability index. The lower the number, the better the stability and the lower the fluctuation.

CONTACTS AND LOCATIONS:
Locations (1):
- Lithuanian Sports University, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No